CLINICAL TRIAL: NCT07294365
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of DZD8586 in Adults With Primary Immune Thrombocytopenia (ITP)
Brief Title: A Study of DZD8586 in Adults With Primary Immune Thrombocytopenia (ITP) (TAI-SHAN11)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZ2025B0002
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DZD8586 dose level 1 (Experimental): Administered orally, once daily.
  Interventions: Drug: DZD8586 dose level 1
- DZD8586 dose level 2 (Experimental): Administered orally, once daily.
  Interventions: Drug: DZD8586 dose level 2
- DZD8586 dose level 3 (Experimental): Administered orally, once daily.
  Interventions: Drug: DZD8586 dose level 3

INTERVENTIONS:
Drug: DZD8586 dose level 1 — DZD8586 will be administered orally in a 28-day cycle.
  Other Names: Birelentinib
  Arms: DZD8586 dose level 1
Drug: DZD8586 dose level 2 — DZD8586 will be administered orally in a 28-day cycle.
  Other Names: Birelentinib
  Arms: DZD8586 dose level 2
Drug: DZD8586 dose level 3 — DZD8586 will be administered orally in a 28-day cycle.
  Other Names: Birelentinib
  Arms: DZD8586 dose level 3

SUMMARY:
This is a Phase 2, open-label, randomized, multicenter study to assess the efficacy and safety of DZD8586 in patients with primary immune thrombocytopenia (ITP). The target population of this study is patients with primary ITP who had failed to respond or relapsed after receiving at least one standard therapy. Participants who meet the inclusion criteria and do not meet the exclusion criteria will be randomized to different dose groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥ 18 years of age.
2. Diagnosed with persistent or chronic primary ITP, and an average of two platelet counts < 30 × 10⁹/L.
3. Have failed at least one standard treatment for ITP (glucocorticoids and/or IVIG).
4. Adequate bone marrow reserve and organ functions.
5. Willing to comply with contraceptive restrictions.

Exclusion Criteria:

1. Have evidence of secondary causes of immune thrombocytopenia.
2. Have a history of coagulation disorders other than ITP, such as disseminated intravascular coagulation, hemolytic uremic syndrome, or thrombotic thrombocytopenic purpura.
3. Any of previous or current treatment prohibited by protocol.
4. Any of severe cardiac abnormalities.
5. Active infection.
6. Poorly controlled gastrointestinal disorder, inadequate absorption of medication or other systemic diseases.
7. Known allergy to DZD8586 drug excipients or other chemical analogues.
8. Pregnant or breastfeeding female participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (4 weeks) | within 4 weeks
  The proportion of patients with platelet counts ≥ 50 × 10⁹/L on 2 consecutive visits (with an interval of at least 7 days) within 4 weeks.

SECONDARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) | 30 days after the last dose
  Safety profiles, for example, adverse events (AEs), serious adverse events (SAEs), ≥ Grade 3 AEs, etc., per Common Terminology Criteria in Adverse Events (CTCAE).
Overall response rate (12 weeks) | within 12 weeks
  The proportion of patients with platelet counts ≥ 50 × 10⁹/L on 2 consecutive visits (with an interval of at least 7 days) within 12 weeks.
Durable response rate | within 24 weeks
  The proportion of patients with platelet counts ≥ 50 × 10⁹/L on at least four of six visits between weeks 14 and 24.
Time to response | within 24 weeks
  Time to first platelet counts ≥ 50 × 10⁹/L.

CONTACTS AND LOCATIONS:
Overall Officials: Hou, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No